CLINICAL TRIAL: NCT04760626
Title: Effectiveness and Safety of Once Weekly Insulin Icodec Used With DoseGuide Versus Once Daily Basal Insulin Analogues in an Insulin naïve Type 2 Diabetes Population in a Clinical Practice Setting
Brief Title: A Research Study to Compare a New Weekly Insulin, Insulin Icodec Used With DoseGuide App, and Daily Insulins in People With Type 2 Diabetes Who Have Not Used Insulin Before
Acronym: ONWARDS 5
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1436-4481; U1111-1247-5279 (Other: World Health Organization (WHO)); 2020-000476-38 (EudraCT Number)
Record Dates: First submitted 2021-02-17; First posted 2021-02-18 (Actual); Results first posted 2025-08-26 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin icodec; Insulin Glargine; insulin degludec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Insulin icodec with DoseGuide (Experimental): Participants randomised to insulin icodec will use insulin icodec with the DoseGuide App to guide their titration.
  Interventions: Drug: Insulin icodec
- Once daily basal insulin analogues (Active Comparator): Participants randomised to basal insulin analogue injections once daily
  Interventions: Drug: Insulin Glargine 100U/mL; Drug: Insulin Degludec; Drug: Insulin Glargine 300U/mL

INTERVENTIONS:
Drug: Insulin icodec — Participants will receive subcutaneous (s.c.) injections of insulin icodec once weekly for 52 weeks.
  Arms: Insulin icodec with DoseGuide
Drug: Insulin Glargine 100U/mL — Participants will receive subcutaneous (s.c.) injections of insulin analogues once daily for 52 weeks.
  Arms: Once daily basal insulin analogues
Drug: Insulin Degludec — Participants will receive subcutaneous (s.c.) injections of insulin analogues once daily for 52 weeks.
  Arms: Once daily basal insulin analogues
Drug: Insulin Glargine 300U/mL — Participants will receive subcutaneous (s.c.) injections of insulin analogues once daily for 52 weeks.
  Arms: Once daily basal insulin analogues

SUMMARY:
This study compares insulin icodec to different daily insulins in people with type 2 diabetes.

The study will look at how well insulin icodec taken once weekly controls blood sugar compared to the insulins taken once daily. Participants will either get insulin icodec, that participants will have to inject once a week on the same day of the week, or a marketed insulin, that participants will have to inject once a day. Which treatment participants get is decided at random.

The insulin is injected with a needle in a skin fold in the thigh, upper arm or stomach.

Participants will measure their blood sugar every day. Participants will get a study phone to record safety data in the electronic diary (eDiary). If participants get a daily insulin they will record their insulin doses in the eDiary. If Participants get weekly insulin icodec, participants study phone will also have the DoseGuide App. The DoseGuide App gives dose recommendations based on their blood sugar and previous doses. Participants will record their insulin doses in the DoseGuide App.

The study will last for about 1 year and 2 months. Participants will have 8 planned clinic visits with the study doctor. More visits will be planned to meet individual needs. At 6 clinic visits participants will have blood samples taken.

Women cannot take part if pregnant, breast-feeding or plan to become pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial.
* Male or female.
* Age above or equal to 18 years at the time of signing informed consent.
* Diagnosed with T2D greater than or equal to 180 days prior to the day of screening.
* HbA1c above 7.0% (53 mmol/mol) as measured by central lab.
* Insulin naïve. However, short term insulin treatment for a maximum of 14 days prior to the day of screening is allowed, as is prior insulin treatment for gestational diabetes.
* Stable daily dose(s) greater than or equal to 90 days prior to the day of screening of any of the following antidiabetic drug(s) or combination regimen(s): a .Any metformin formulations greater than or equal to 1500 mg or maximum tolerated or effective dose. b .Any metformin combination formulations greater than or equal to 1500 mg or maximum tolerated or effective dose. c. Any of the following non-insulin antidiabetic drug classes including combinations (greater than or equal to half of the maximum approved dose according to local label or maximum tolerated or effective dose):i). Sulfonylureas ii). Meglitinides (glinides) iii). DPP-4 inhibitors iv. SGLT2 inhibitors v). Thiazolidinediones vi). Alpha-glucosidase inhibitors vii). Oral combination products (for the allowed individual Oral Antidiabetic Drugs (OADs)) viii). Oral or injectable GLP-1-receptor agonists.
* Intensification with insulin is indicated to achieve glycaemic target (4.4-7.2 mmol/L, 80-130 mg/dL) at the discretion of the treating investigator.

Exclusion Criteria:

* Known or suspected hypersensitivity to trial product(s) or related products.
* Previous participation in this trial. Participation is defined as signed informed consent.
* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate contraceptive method (adequate contraceptive measures as required by local regulation or practice).
* Participation in any clinical trial of an approved or non-approved investigational medicinal product within 30 days before screening. (Simultaneous participation in a trial with the primary objective of evaluating an approved or non-approved investigational medicinal product for prevention or treatment of COVID-19 disease or postinfectious conditions is allowed if the last dose of the investigational medicinal product has been received more than 30 days before screening)
* Any disorder which in the investigator's opinion might jeopardise subject's safety.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1085 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2022-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (180):
- United States (79):
  - Univ of Alabama Birmingham, Birmingham, Alabama
  - Lakeview Clinical Research, LLC, Guntersville, Alabama
  - American Clinical Trials, Buena Park, California
  - San Fernando Valley Hlth Inst, LLC, Canoga Park, California
  - Valley Research, Fresno, California
  - Advanced Investigative Medicine, Inc., Hawthorne, California
  - Diabetes/Lipid Mgmt & Res Ctr, Huntington Beach, California
  - Scripps Whittier Diabetes Inst, La Jolla, California
  - First Valley Medical Group, Lancaster, California
  - Torrance Clin Res Inst, Inc., Lomita, California
  - Valley Clinical Trials, Inc., Northridge, California
  - Desert Oasis Hlthcr Med Group, Palm Springs, California
  - Clinical Trials Research_Sacramento, Sacramento, California
  - San Diego Family Care, San Diego, California
  - NorCal Endocrinology and Internal Medicine, San Ramon, California
  - Encompass Clinical Research_Spring Valley, Spring Valley, California
  - Coastal Metabolic Research Center, Ventura, California
  - Est Cst Inst for Rsrch,Jksnvil, Jacksonville, Florida
  - Adult Medicine of Lake County, Inc., Mt. Dora, Florida
  - Suncoast Clin Res Port Richey, New Port Richey, Florida
  - Florida Inst For Clin Res, Orlando, Florida
  - Palm Harbor Medical Associates, Palm Harbor, Florida
  - Suncoast Clinical Research, Inc., Palm Harbor, Florida
  - Metabolic Research Institute Inc, West Palm Beach, Florida
  - Clinical Research of Cent FL, Winter Haven, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Endo Res Solutions, Inc, Roswell, Georgia
  - Elite Clinical Trials, Blackfoot, Idaho
  - Cedar-Crosse Research Center, Chicago, Illinois
  - Central Illinois Diabetes and Clinical Research, Springfield, Illinois
  - Cotton O'Neil Diab & Endo Ctr, Topeka, Kansas
  - MedStar Community Clin Res Ctr, Hyattsville, Maryland
  - Endo and Metab Consultants, Rockville, Maryland
  - Northern Pines Hlth Ctr, PC, Buckley, Michigan
  - Arcturus Healthcare, PLC., Troy, Michigan
  - Jefferson City Medical Group, PC, Jefferson City, Missouri
  - Methodist Physicians Clin, Omaha, Nebraska
  - Univ of Nebraska Medical CTR, Omaha, Nebraska
  - Palm Research Center Inc-Vegas, Las Vegas, Nevada
  - Southern New Hampshire Diabetes and Endocrinology, Nashua, New Hampshire
  - Albuquerque Clin Trials, Inc., Albuquerque, New Mexico
  - AMC Community Endocrinology, Albany, New York
  - N.Y. Total Medical Care PC, Brooklyn, New York
  - Mid Hudson Medical Research, PLLC, New Windsor, New York
  - Endocrine Associates of Long Island, PC, Smithtown, New York
  - Southgate Medical Group, LLP, West Seneca, New York
  - Physicians East Endocrinology, Greenville, North Carolina
  - Medication Management, LLC, Raleigh, North Carolina
  - Accellacare, Wilmington, North Carolina
  - Plains Clinical Research Center, LLC_Fargo, Fargo, North Dakota
  - Diab & Endo Assoc of Stark Co, Canton, Ohio
  - Providence Health Partners Ctr, Dayton, Ohio
  - New Venture Medical Research, Wadsworth, Ohio
  - The Diabetes Center, LLC, Murrells Inlet, South Carolina
  - Hillcrest Clinical Research, Simpsonville, South Carolina
  - AM Diabetes And Endocrinology Center, Bartlett, Tennessee
  - Chattanooga Medical Research, LLC, Chattanooga, Tennessee
  - Univ Diab & Endo Consultants, Chattanooga, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - HealthStar Physicians PC, Morristown, Tennessee
  - Amarillo Med Spec LLP, Amarillo, Texas
  - Texas Diab & Endo, P.A., Austin, Texas
  - Texas Diabetes & Endocrinology, Austin, Texas
  - Velocity Clinical Res-Dallas, Dallas, Texas
  - UT Southwestern Med Cntr, Dallas, Texas
  - PrimeCare Medical Group, Houston, Texas
  - Juno Research, LLC, Houston, Texas
  - Protenium Clinical Research, Hurst, Texas
  - Medical Colleagues-Texas LLP, Katy, Texas
  - Fmc Science, Llc, Lampasas, Texas
  - Andres Garcia-Zuniga, MD, P.A, Laredo, Texas
  - Texas Diab & Endo, P.A., Round Rock, Texas
  - Clinical Trials of Texas, LLC, San Antonio, Texas
  - NE Clin Res of San Antonio, San Antonio, Texas
  - Simcare Medical Research, LLC, Sugar Land, Texas
  - Wade Family Medicine, Bountiful, Utah
  - Chrysalis Clinical Research, St. George, Utah
  - TPMG Clinical Research, Newport News, Virginia
  - Clinical Inv Spec, Inc.Kenosha, Kenosha, Wisconsin
- Canada (35):
  - LMC Clin Res Inc. Calgary, Calgary, Alberta
  - The Bailey Clinic, Red Deer, Alberta
  - Dr. M.B. Jones Inc, Victoria, British Columbia
  - Rivergrove Medical Clinic, Winnipeg, Manitoba
  - Winnipeg Clinic, Winnipeg, Manitoba
  - G.A. Research Associates Ltd., Moncton, New Brunswick
  - Commonwealth Medical Clinic, Mount Pearl, Newfoundland and Labrador
  - Eastern Health Authority, St. John's, Newfoundland and Labrador
  - LMC Diabetes & Endocrinology (Barrie), Barrie, Ontario
  - Centricity Research LMC, Brampton, Ontario
  - LMC Clinical Res Thornhill, Concord, Ontario
  - Medical Trust Clinics, Inc., Courtice, Ontario
  - LMC Endo Ctr (Etobicoke) Ltd, Etobicoke, Ontario
  - Wharton Med Clin Trials, Hamilton, Ontario
  - Premier Clinical Trial Research Network (PCTRN), Hamilton, Ontario
  - Milestone Research, London, Ontario
  - Western Univ. Cnt for Studies in Fam Med, London, Ontario
  - LMC Research Inc. Ottawa, Nepean, Ontario
  - LMC Oakville, Oakville, Ontario
  - Bluewater Clin Res Group,Inc, Sarnia, Ontario
  - Winterberry Family Medicine, Stoney Creek, Ontario
  - LMC Endo Centres Ltd.(Bayview), Toronto, Ontario
  - Dr. Anil K Gupta Medicine Professional Corporation, Toronto, Ontario
  - ViaCar Recherche Clinique Inc, Brossard, Quebec
  - Ecogene-21, Chicoutimi, Quebec
  - Ctr de rech Clin de Laval, Laval, Quebec
  - Manna Research Mirabel, Mirabel, Quebec
  - Applied Med Inf Res, Montreal, Quebec
  - Diex Recherche Joliette, Saint-Charles-Borromée, Quebec
  - LMC Clin Rsrch Inc. (Montreal), Saint-Laurent, Quebec
  - Ctr Méd. et pro d l'Ost d port, Saint-Marc-des-Carrieres, Quebec
  - Diex Recherche Victoriaville, Victoriaville, Quebec
  - Recherche Clinique Sigma inc, Québec
  - Diex Recherche Quebec Inc., Québec
  - Centre de Recherche Saint-Louis, Québec
- Germany (14):
  - Diabetespraxis Mergentheim, Bad Mergentheim
  - Medizinisches Versorgungszentrum Am Bahnhof Spandau GbR, Berlin
  - InnoDiab Forschung GmbH, Essen
  - Zentrum für klinische Forschung, Dr. med. Lüdemann, Falkensee
  - Wendisch/Dahl Hamburg (DZHW), Hamburg
  - Milek, Hohenmölsen, Hohenmölsen
  - Institut für Diabetesforschung GmbH Münster - Dr. med. Rose, Münster
  - MedicalCenter am Clemenshospital - Schwerpunktpraxis für Diabetologie und Ernährungsmedizin, Münster
  - RED-Institut für medizinische Forschung und Fortbildung GmbH, Oldenburg in Holstein
  - Praxis Dr. med. Wenzl-Bauer, Rehlingen-Siersburg
  - Med.Versorgungszentrum Riesa-Dr. Bieler, Riesa
  - Zentrum für klinische Studien Alexander Segner, Saint Ingbert-Oberwürzbach
  - MZM Praxis Drs. Erlinger, Stuttgart
  - Zentrum für klinische Studien Allgäu Oberschwaben, Wangen
- Greece (13):
  - Iatriko Psychicou Private Clinic, Athens
  - 'G. Gennimatas' General Hospital of Athens, Athens
  - "Laiko" General Hospital of Athens, Athens
  - Iatriko Athinon 'Palaiou Falirou', Athens
  - Korgiallenio - Benakio Hospital (Red Cross Hosp.), Athens
  - Univ Gen Hospital Larisa, Larissa
  - General Hospital of Thessaloniki 'G. Gennimatas, Thessaloniki
  - AHEPA General University Hospital, Thessaloniki
  - "Ippokrateio" G.H. of Thessaloniki, Thessaloniki
  - EUROMEDICA Gen Clinic The/ki, Endocrin,Metabolism,Diabetes, Thessaloniki
  - "Thermi" Private Hosital, Thessaloniki
  - General Hospital of Thessaloniki "G.Papanikolaou", Thessaloniki
  - "Ippokrateio" General Hosp Thessaloniki, A' Internal Med, Thessaloniki
- Hungary (13):
  - Belinus Bt., Debrecen, Hajdú-Bihar
  - Komáromi Selye János Kórház, Komárom, Komárom-Esztergom
  - Szent Margit Kórház, Budapest
  - Óbudai Egészségügyi Centrum, Budapest
  - Szőcs Depot Egészségügyi Szolgáltató Kft., Budapest
  - ClinDiab Egészségügyi Szolgáltató és Kereskedelmi Kft., Budapest
  - MED-TIMA Kft., Budapest
  - MH Egészségügyi Központ, Budapest
  - Uno Medical Trials Eü. Szolgáltató és Kereskedelmi Kft., Budapest
  - Kaposi Mór Oktató Kórház, Kaposvár
  - Szegedi Tudomanyegyetem St Györgyi Albert Klinikai Központ, Szeged
  - Vas Vármegyei Markusovszky Egyetemi Oktatókórház, Szombathely
  - Zala Megyei Szent Rafael Kórház, Zalaegerszeg
- Poland (11):
  - Centrum Medyczne Pratia Gdynia, Gdynia, Pomeranian Voivodeship
  - NZOZ Gdanska Poradnia Cukrzycowa Sp.z o.o., Gdansk
  - Centrum Medyczne Pratia Katowice, Katowice
  - Gabinet Lekarski Malgorzata Saryusz-Wolska, Lodz
  - Pro Salus Centrum Medyczne, Lodz
  - Katedra i Klinika Chorob Wewnetrznych AM w Lublinie, Lublin
  - Oddzial Chorób - Wewn., Poznan
  - Velocity Nova Sp. z o.o., Puławy
  - Lubelskie Centrum Diagnostyczne Tomasz Blicharski, Świdnik
  - Poradnia dla Chorych na Cukrzycę, Zabrze
  - Velocity Nova Sp. z o.o., Staszów, Świętokrzyskie Voivodeship
- Manati Ctr For Clin Research, Manatí, Puerto Rico
- Turkey (Türkiye) (14):
  - T.C. Saglık Bakanlıgı Adana Sehir Egitim ve Arastirma Hastan, Adana
  - Baskent Universitesi Adana, Adana
  - Ankara Universitesi Ibni Sina Hastanesi, Ankara
  - Gaziantep Universitesi Tip Fakultesi Hastanesi, Gaziantep
  - Hatay Mustafa Kemal Universitesi Saglik Uygulama ve Arastirm, Hatay
  - Kanuni Sultan Suleyman Egitim ve Arastirma Hastanesi, Istanbul
  - Seyrantepe Hamidiye Etfal Egitim ve Arastirma Hastanesi, Istanbul
  - Istanbul Universitesi Istanbul Tip Fakultesi - Endokrinoloji, Istanbul
  - Haydarpasa Numune Hastanesi, Istanbul
  - T.C SB Goztepe Prof. Dr. Suleyman Yalcin City Hospital, Istanbul
  - Umraniye Egitim ve Arastirma Hastanesi, Istanbul
  - T.C. S.B. Ist Il SagMud Pendik Egitim ve Arastirma Hastanesi, Istanbul
  - Dokuz Eylul University Medical Faculty, Izmir
  - Erciyes Universitesi Tip Fakultesi, Kayseri

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Result] Philis-Tsimikas A, Bajaj HS, Begtrup K, Cailleteau R, Gowda A, Lingvay I, Mathieu C, Russell-Jones D, Rosenstock J. Rationale and design of the phase 3a development programme (ONWARDS 1-6 trials) investigating once-weekly insulin icodec in diabetes. Diabetes Obes Metab. 2023 Feb;25(2):331-341. doi: 10.1111/dom.14871. Epub 2022 Oct 14. PMID 36106652
- [Derived] Philis-Tsimikas A, Krogsdahl Bache J, Fu A, Kellerer M, Salvesen-Sykes K, Bain SC. Insights on Hospitalisations from the Phase 3a ONWARDS 1-6 Trials of Once-Weekly Insulin Icodec. Diabetes Ther. 2025 Aug;16(8):1615-1631. doi: 10.1007/s13300-025-01745-4. Epub 2025 Jun 4. PMID 40465144
- [Derived] Riddell MC, Heller S, Carstensen L, Rocha TMP, Kehlet Watt S, Woo VC. The effect of once-weekly insulin icodec vs once-daily basal insulin on physical activity-attributed hypoglycaemia in type 2 diabetes: a post hoc analysis of ONWARDS 1-5. Diabetologia. 2025 Jul;68(7):1416-1422. doi: 10.1007/s00125-025-06414-6. Epub 2025 Apr 5. PMID 40186685
- [Derived] Billings LK, Asong M, Bog M, Clancy S, Kruse C, de Laguiche E, Maddaloni E. AUGMENTed Real-World Data Enhances Comparative Efficacy Between Once-Weekly Insulin Icodec with Dosing Guide App Versus Once-Daily Insulin Glargine U300 in Insulin-Naive Type 2 Diabetes. Diabetes Ther. 2025 Feb;16(2):227-239. doi: 10.1007/s13300-024-01679-3. Epub 2024 Dec 19. PMID 39699848
- [Derived] Polonsky W, Benamar M, Carstensen L, Davies M, Meller Donatsky A, Franek E, Kellerer M, Philis-Tsimikas A, Goldenberg R. Improved treatment satisfaction with once-weekly insulin icodec compared with once-daily basal insulin in individuals with type 2 diabetes: An analysis of patient-reported outcomes and participant interviews from ONWARDS 2 and 5 and a physician survey from ONWARDS 1. Diabetes Res Clin Pract. 2024 Nov;217:111885. doi: 10.1016/j.diabres.2024.111885. Epub 2024 Oct 4. PMID 39368488
- [Derived] Bajaj HS, Aberle J, Davies M, Donatsky AM, Frederiksen M, Yavuz DG, Gowda A, Lingvay I, Bode B. Once-Weekly Insulin Icodec With Dosing Guide App Versus Once-Daily Basal Insulin Analogues in Insulin-Naive Type 2 Diabetes (ONWARDS 5) : A Randomized Trial. Ann Intern Med. 2023 Nov;176(11):1476-1485. doi: 10.7326/M23-1288. Epub 2023 Sep 26. PMID 37748181

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 182 sites in Canada, Germany, Greece, Hungary, Poland, Turkey and the United States.
Groups:
- Insulin Icodec: Participants were to receive once weekly subcutaneous (s.c.) injection of Insulin icodec guided by the DoseGuide app, for 52 weeks using PDS290 prefilled pen-injector. Participants were to perform once daily pre-breakfast self-monitoring plasma glucose (SMPG). The dose was adjusted based on 3 pre-breakfast SMPG values measured on the 2 previous days and the day of the contact. If at least one pre-breakfast SMPG value was: lesser than (<) 4.4 millimoles per liter (mmol/L): dose reduced by 20 units (U); 4.4-7.2 mmol/L: no adjustment; greater than (>) 7.2 mmol/L: dose increased by 20 U.
- Once Daily Basal Insulin Analogue: Participants were to receive once daily basal insulin analogue of (Insulin degludec using PDS290 prefilled pen-injector) or (Insulin glargine U100 or Insulin glargine U300 using SoloSTAR® pre-filled pen-injector) for 52 weeks, at a dose in accordance with local label. Titration of once daily basal insulin analogue comparators is at the discretion of the investigator according to local clinical practice. The recommended doses for all once daily basal insulin analogues was based on the locally approved label.
Period: Overall Study
Arm/Group | Insulin Icodec | Once Daily Basal Insulin Analogue
Started | 542 | 543
Full Analysis Set (FAS) | 542 | 543
Safety Analysis Set (SAS) | 542 | 538
Completed | 497 | 493
Not Completed | 45 | 50
Not completed — Withdrawal by Subject | 24 | 20
Not completed — Lost to Follow-up | 14 | 19
Not completed — Physician Decision | 3 | 5
Not completed — Death | 3 | 6
Not completed — Site closure | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set included all randomised participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Icodec | Once Daily Basal Insulin Analogue | Total
Number analyzed (Participants) | 542 | 543 | 1085
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.15 (10.79) | 59.39 (10.15) | 59.27 (10.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 233 | 230 | 463
  Male | 309 | 313 | 622
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 51 | 44 | 95
  Not Hispanic or Latino | 490 | 499 | 989
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian Or Alaska Native | 2 | 1 | 3
  Asian | 28 | 19 | 47
  Black Or African American | 24 | 28 | 52
  Native Hawaiian Or Other Pacific Islander | 2 | 1 | 3
  Not Reported | 1 | 0 | 1
  White | 478 | 493 | 971
  Other | 7 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycated Haemoglobin (HbA1c)
Description: Change in HbA1c from baseline (week 0) to week 52 is presented.
Time Frame: Baseline (week 0), week 52
Population: Full analysis set included all randomised participants. Overall number of participants analyzed = participants with available data for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | Insulin Icodec | Once Daily Basal Insulin Analogue
Number analyzed (Participants) | 542 | 542
Percentage of HbA1c | -1.68 (0.09) | -1.31 (0.12)
Statistical Analysis 1: Comparison: Insulin Icodec vs Once Daily Basal Insulin Analogue; The response and change from baseline in response after 52 weeks were analysed using an analysis of covariance (ANCOVA) model with region and randomised treatment as fixed factors, and baseline HbA1c as a covariate; Test type: Non-Inferiority — Non-inferiority of insulin icodec was considered confirmed if the upper limit of the two-sided 95% confidence interval (CI) for mean treatment difference (insulin icodec with doseguide minus once daily basal insulin analogue) was strictly below 0.3 percent point; p < 0.0001, ANCOVA; Treatment difference = -0.38, 95% CI 2-sided [-0.66 to -0.09]

2. Secondary Outcome: Time From Baseline to Treatment Discontinuation or Intensification
Description: Time from baseline to treatment discontinuation or intensification from baseline (week 0) to week 52 is presented.
Time Frame: From baseline (week 0) to week 52
Population: FAS included all randomised participants. Overall number of participants analyzed = participants with available data for this outcome measure.
Measure: Median (Full Range); unit: Weeks
Arm/Group | Insulin Icodec | Once Daily Basal Insulin Analogue
Number analyzed (Participants) | 59 | 50
Weeks | 20.1 [0.0 to 51.0] | 13.9 [0.0 to 55.1]

3. Secondary Outcome: Change in Diabetes Treatment Satisfaction Questionnaire (DTSQs) in Total Treatment Satisfaction
Description: Change in DTSQs in total treatment satisfaction is presented. The DTSQs questionnaire was used to assess participants treatment satisfaction which contained 8 components (DTSQs Item 1-8 : how satisfied are you with your current treatment, how often have you felt that blood sugars have been unacceptably high, how often have you felt that blood sugars have been unacceptably low, how convenient have you been finding your treatment to be recently, how flexible have you been finding your treatment to be recently, how satisfied are you with your understanding of your diabetes, would you recommend treatment to someone else with your kind of diabetes, how satisfied would you be to continue with present form of treatment). The result presented is the treatment satisfaction summary score, which is the sum of 6 of the 8 items of the DTSQs questionnaire. Total scores for treatment satisfaction range from 0-36 with 0 being the lowest and 36 being the highest score in total treatment satisfaction.
Time Frame: Baseline (week 0), week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Insulin Icodec | Once Daily Basal Insulin Analogue
Number analyzed (Participants) | 513 | 500
Score on a scale | 4.68 (0.25) | 3.90 (0.25)

4. Secondary Outcome: Treatment Related Impact Measure for Diabetes (TRIM-D) Compliance Domain
Description: Treatment Related Impact Measure for Diabetes (TRIM-D) Compliance domain at week 52 is presented. The TRIM-D questionnaire was developed to capture the impact of diabetes treatment on patients' functioning and well-being. The questionnaire was used to measure the compliance between the treatment groups. The total TRIM-D compliance score is computed by summing across the items and then transforming to a 0-100 scale with higher score indicating better compliance.
Time Frame: At end of treatment (week 52)
Population: FAS included all randomised subjects.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Insulin Icodec | Once Daily Basal Insulin Analogue
Number analyzed (Participants) | 542 | 543
Score on a scale | 90.42 (0.64) | 87.37 (0.64)

5. Secondary Outcome: Number of Severe Hypoglycaemic Episodes (Level 3)
Description: Number of severe hypoglycaemic episodes (level 3) is presented. Severe hypoglycaemia (level 3) is defined as hypoglycaemia with severe cognitive impairment requiring external assistance for recovery.
Time Frame: From baseline (week 0) to week 57
Population: Safety analysis set included all participants who were randomly assigned to trial treatment and who took at least 1 dose of trial product. Overall number of participants analyzed = participants with available data for this outcome measure.
Measure: Number; unit: Episodes
Arm/Group | Insulin Icodec | Once Daily Basal Insulin Analogue
Number analyzed (Participants) | 542 | 538
Episodes | 0 | 5

6. Secondary Outcome: Number of Clinically Significant Hypoglycaemic Episodes (Level 2) (Below 3.0 Millimoles Per Liter [mmol/L] (54 Milligrams Per Deciliter [mg/dL]), Confirmed by Blood Glucose (BG) Meter)
Description: Number of clinically significant hypoglycaemic episodes (level 2) (below 3.0 millimoles per liter [mmol/L] (54 mg/dL), confirmed by BG meter) is presented. Clinically significant hypoglycaemia (level 2) is defined as plasma glucose value of less than (<) 3.0 mmol/L (54 mg/dL) confirmed by BG meter.
Time Frame: From baseline (week 0) to week 57
Population: as for outcome 5
Measure: Number; unit: Episodes
Arm/Group | Insulin Icodec | Once Daily Basal Insulin Analogue
Number analyzed (Participants) | 542 | 538
Episodes | 104 | 76

7. Secondary Outcome: Number of Clinically Significant Hypoglycaemic Episodes (Level 2) (Below 3.0 mmol/L (54 mg/dL), Confirmed by BG Meter) or Severe Hypoglycaemic Episodes (Level 3)
Description: Number of clinically significant hypoglycaemic episodes (level 2) (below 3.0 mmol/L (54 mg/dL), confirmed by BG meter) or severe hypoglycaemic episodes (level 3) is presented. Clinically significant hypoglycaemia (level 2) is defined as plasma glucose value of less than (<) 3.0 mmol/L (54 mg/dL) confirmed by BG meter. Severe hypoglycaemia (level 3) is defined as hypoglycaemia with severe cognitive impairment requiring external assistance for recovery.
Time Frame: From baseline (week 0) to week 57
Population: as for outcome 5
Measure: Number; unit: Episodes
Arm/Group | Insulin Icodec | Once Daily Basal Insulin Analogue
Number analyzed (Participants) | 542 | 538
Episodes | 104 | 81

ADVERSE EVENTS:
Time Frame: From baseline week 0 to week 57
Description: All presented AEs are treatment emergent. Treatment emergent adverse events (TEAEs): events that had onset date during on-treatment period, time period in which participants was considered exposed to trial product. Safety analysis set included all randomised participants randomly assigned to trial treatment who took at least 1 dose of trial product. AEs were assessed in SAS and All-Cause Mortality was assessed for all enrolled participants.
Arm/Group | Insulin Icodec | Once Daily Basal Insulin Analogue
All-Cause Mortality (participants affected / at risk) | 3/542 | 6/543
Serious Adverse Events (participants affected / at risk) | 45/542 | 57/538
Other Adverse Events (participants affected / at risk) | 43/542 | 55/538
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Icodec (N=542) | Once Daily Basal Insulin Analogue (N=538)
Acute coronary syndrome (Cardiac disorders) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 3 (3)
Acute myocardial infarction (Cardiac disorders) | 4 (4) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1)
Arrhythmia (Cardiac disorders) | 2 (2) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 3 (3) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 3 (3)
Cardiac arrest (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure (Cardiac disorders) | 3 (3) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac pacemaker replacement (Surgical and medical procedures) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Cerebral artery embolism (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral atrophy (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Cholecystitis infective (Infections and infestations) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 2 (2) | 5 (5)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Drug intolerance (General disorders) | 1 (1) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Eosinophilic oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Herpes zoster infection neurological (Infections and infestations) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertensive urgency (Vascular disorders) | 0 (0) | 1 (1)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 1 (1) | 0 (0)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Localised oedema (General disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Ocular ischaemic syndrome (Eye disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Periprocedural myocardial infarction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Peritonsillar abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural inflammation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin neoplasm excision (Surgical and medical procedures) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stress urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sweat gland infection (Infections and infestations) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Venous stenosis (Vascular disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
White matter lesion (Nervous system disorders) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Icodec (N=542) | Once Daily Basal Insulin Analogue (N=538)
COVID-19 (Infections and infestations) | 43 (46) | 55 (57)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2020-11-23): https://cdn.clinicaltrials.gov/large-docs/26/NCT04760626/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-14): https://cdn.clinicaltrials.gov/large-docs/26/NCT04760626/SAP_001.pdf